CLINICAL TRIAL: NCT02368847
Title: Optimizing and Validating the Clinical Algorithm for Diagnosing Urinary Tract Infections in Older Persons Admitted to a Psychogeriatric Ward
Brief Title: Urinary Tract Infections in Older Persons Admitted to a Psychogeriatric Ward
Acronym: UTI_UCP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Latour Katrien, Research Assistant, KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UTI_UCP
Record Dates: First submitted 2015-02-09; First posted 2015-02-23 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Urinary Tract Infections
Keywords: Aged; Psychiatric Hospitals
MeSH Terms: conditions — Urinary Tract Infections | interventions — Diagnostic Tests, Routine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diagnostic tests (Other): For any patient with a suspected urinary tract infection during the course of the study a basic questionnaire will have to be filled out and diagnostic tests (urine sample for culture, dipstick assay for the detection of nitrites and leukocyte- esterase and a POC CRP test) will have to be perform.
  Interventions: Device: Diagnostic tests

INTERVENTIONS:
Device: Diagnostic tests — C Reactive Protein (CRP) measurement on capillary blood using a point-of-care test to determine C Reactive Protein level in the blood
Device: Diagnostic tests — Uricult dipslide: Easy-to-perform bacterial culture test for dectecting urinary tract infections in point of care settings

SUMMARY:
Urinary tract infections are one of the most common types of infections in older persons. The general aim of this study is to improve the epidemiological knowledge and develop a better diagnostic algorithm for urinary tract infections in older institutionalized individuals in order to reduce excessive prescribing of antibiotics and prevent antimicrobial resistance.

ELIGIBILITY:
Inclusion Criteria:

* Older (65+ years) persons admitted to a gerontopsychiatric ward

Exclusion Criteria:

* Patients not understanding Dutch or not willing to participate (no informed consent)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-03; Primary Completion 2015-08 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Serious infection | 2 months
  To verify if the elderly has a serious infection, the research team will combine test results (dipstick, dipslide and CRP measurement) with signs/symptoms reported in the patient questionnaire.

SECONDARY OUTCOMES:
Reliability of the uricult dipslide in a population of institutionalized older patients | 2 months
  To verify the reliability of the uricult dipslide, a comparison will be made between the result of a dipslide read after 48h at room temperature, a dipslide incubated for 24h at +/- 35° Celsius and a urine culture test performed in a microbiology lab

CONTACTS AND LOCATIONS:
Overall Officials: Jan De Lepeleire, PhD, Study Director — KU Leuven